CLINICAL TRIAL: NCT05484791
Title: Acute Effect Of The Lumbar Rotational Spinal Mobilization Technique On Pain, Disability And Radiological Findings Of Patients With Lumbar Disc Herniation
Brief Title: The Effect of a Lumbar Rotational Spinal Mobilization Technique With Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01/10/2019-E.13568
Record Dates: First submitted 2022-07-19; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar disc herniation; Manual therapy; Lumbar Spinal Rotational Mobilization
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: The research was designed as a semi-experimental study with pre-test (before implementation), post-test (after implementation) and 2-month follow-up assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Lumbar Rotational Spinal Mobilization Technique (Experimental): Patients included in the study underwent the lumbar rotational spinal mobilization technique during two sessions per week
  Interventions: Other: The Lumbar Rotational Spinal Mobilization Technique

INTERVENTIONS:
Other: The Lumbar Rotational Spinal Mobilization Technique — Patients included in the study underwent the lumbar rotational spinal mobilization(LRSM) technique during two sessions per week. The LRSM technique is applied while patients are lying on their side. The uppermost hip and knee are placed in 90 degree flexion, this is to assist rotational stress, and the lower leg is placed in extension. The lower shoulder is strongly pulled; thus, the upper shoulder is positioned toward the posterior and the pelvis moves anteriorly. The clinician stands in front of the patient. They stabilize the upper shoulder with one hand, and place the palm of the other hand behind the hard part of the ilium wing, with forearm horizontal and fingers turned toward the clinician. A rotational force is applied with pressure in the horizontal direction by pulling the hand on the ilium toward the clinician. In this position, 30 slow repeated movements are performed. The same practice is performed on both sides

SUMMARY:
The aim of this study was to research the effect of the Lumbar Spinal Rotational Mobilization technique on radiological findings, pain, disability and joint range of motion (ROM) in patients with lumbar disc herniation

DETAILED DESCRIPTION:
In our study, it was aimed to investigate the acute effect of Lumbar Rotational Spinal Mobilization Technique on radiological findings, pain, disability and range of motion in 26 patients diagnosed with lumbar disc herniation(LDH) by magnetic resonance imaging(MRI) and physical examination. Disc height, herniation distance and facet joint distance of the patients were measured with MRI. Pain was assessed with the Visual Analogue Scale. Disability was measured with the Oswestry Low Back Pain Disability Questionnaire and Lumbar range of motion(ROM) was measured with a goniometer and tape measure. Rotational Spinal Mobilization Technique was applied to the patients in 2 sessions with a one-week interval, slowly and with 30 repetitions in both directions. All assessments were repeated within 1 week after treatment. It was observed whether there was an improvement in terms of radiological, pain, disability and ROM in the patients. 2 months after the 2nd evaluation, other parameters except the radiological evaluation were reapplied and it was tried to determine whether the effect persisted.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with LDH by MRI and physical examination
* Having pain due to LDH
* Be between the ages of 18 and 65

Exclusion Criteria:

* History Of Spinal Surgery
* History Of Autoimmune Disease (Ankylosing Spondylitis, Rheumatoid Arthritis Or Other Disease)
* Spondylolysis Or Spondylolisthesis
* Spinal Fracture
* Cardiac Pathology
* Stroke History
* Cauda Equina Syndrome,
* Continuous Painkiller Drug Use
* Spinal inflammation
* Spinal Tumor
* Corticosteroid Drug Use İn The Last Month
* Osteoporosis

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Assessing disc height change | Disc height, was measured twice by a radiology expert 1 week before and 1 week after treatment
  Images for radiological assessment of patients were obtained with a 1.5 Tesla GE brand Magnetic Resonance (MR) device. Sagittal T2A and axial T2A sequences were used. If the same person had herniation at different levels, the level with highest degree of herniation was included in the assessment. All MR images were obtained during the day between 16:00 and 18:00 hours
Assessing disc herniation thickness change | Disc herniation thickness was measured twice by a radiology expert 1 week before and 1 week after treatment
  Images for radiological assessment of patients were obtained with a 1.5 Tesla GE brand Magnetic Resonance (MR) device. Sagittal T2A and axial T2A sequences were used. If the same person had herniation at different levels, the level with highest degree of herniation was included in the assessment. All MR images were obtained during the day between 16:00 and 18:00 hours
Assessing facet joint distance change | Facet joint distance was measured twice by a radiology expert 1 week before and 1 week after treatment
  Images for radiological assessment of patients were obtained with a 1.5 Tesla GE brand Magnetic Resonance (MR) device. Sagittal T2A and axial T2A sequences were used. If the same person had herniation at different levels, the level with highest degree of herniation was included in the assessment. All MR images were obtained during the day between 16:00 and 18:00 hours

SECONDARY OUTCOMES:
Functional capacity change assessment | The functional capacity of patients participating in the study was assessed 1 week before, 1 week and 2 months after treatment using the Oswestry Low Back Pain Disability Questionnaire.
  The Oswestry Low Back Pain Disability Questionnaire (OLBPDQ) was used to assess disability levels and quality of life linked to low back pain of patients. The OLBPDQ was developed to assess disability linked to pain for people with acute, subacute or chronic low back pain. The OLBPDQ contains 1 item related to pain and 9 items related to daily life activities (personal care, lifting, walking, sitting, standing, sleep, sexual life, social life and travel). Each item is rated on a 6-point scale ranked from the best scenario to the worst scenario. Points for each item increase by 1 for each response choice from 0 (first response choice) to 5 (final response choice). Missing values are skipped. Total points are calculated as a percentage value
Pain change assessment | Pain assessment was recorded 1 week before, 1 week and 2 months after treatment
  The pain levels felt by patients in their low back and surrounding regions was assessed with the visual analog scale (VAS). On this assessment, the patient expresses the pain levels felt by marking their position on a 10 cm scale numbered from 0 to 10 where 0 indicates no pain and 10 indicates unbearable pain. Cases are requested to express their pain by marking the appropriate number for their pain level on the scale and the value is recorded in cm.

OTHER OUTCOMES:
Evaluation of joint range of motion change | Joint range of motion was assessed and recorded 1 week before, 1 week and 2 months after treatment
  All patients participating in the study had lumbar flexion, lumbar extension, lumbar lateral flexion and lumbar rotations measured. Lumber flexion and lumbar lateral flexion were obtained by measuring the distance between the ground and middle finger tip with a tape measure. Lumber extension and lumbar rotations were measured with a goniometer

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Taşkent, Study Chair — Muş State Hospital; Mahmut Çakıllı, Study Chair — Muş State Hospital
Locations (1):
- Muş Alparslan University, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No